CLINICAL TRIAL: NCT03148470
Title: Impact of Theta Burst Stimulation Over the Left Dorsolateral Prefrontal Cortex on Language Switching and Cognitive Flexibility
Brief Title: Impact of Theta Burst Stimulation Over the Left DLPFC on Language Switching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean-Marie Annoni (Other)
Responsible Party: Sponsor-Investigator, Jean-Marie Annoni, Prof. Dr. med., University of Fribourg
Organization: University of Fribourg (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: SNF325130_156937_4
Record Dates: First submitted 2017-05-01; First posted 2017-05-11 (Actual); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Languages
Keywords: theta burst stimulation; Language switching; dorsolateral prefrontal cortex
MeSH Terms: conditions — Language

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intermittent theta burst stimulation (Experimental): intermittent theta burst stimulation (iTBS) + Sham iTBS
  Interventions: Device: Sham iTBS; Device: intermittent theta burst stimulation (iTBS)
- continuous theta burst stimulation (Experimental): continuous theta burst stimulation (cTBS) + Sham cTBS
  Interventions: Device: Sham cTBS; Device: continuous theta burst stimulation (cTBS)

INTERVENTIONS:
Device: Sham iTBS — Placebo stimulation for the iTBS group
  Arms: intermittent theta burst stimulation
Device: Sham cTBS — Placebo stimulation for the cTBS group
  Arms: continuous theta burst stimulation
Device: intermittent theta burst stimulation (iTBS) — Excitatory theta burst stimulation
  Arms: intermittent theta burst stimulation
Device: continuous theta burst stimulation (cTBS) — inhibitory theta burst stimulation
  Arms: continuous theta burst stimulation

SUMMARY:
The purpose of this study is to investigate whether theta burst stimulation (TBS) over the left dorsolateral prefrontal cortex (DLPFC) influences language switching and cognitive flexibility. The experimental paradigm will assess the impact of inhibitory and excitatory prefrontal stimulation by TBS versus sham-TBS over the DLPFC in healthy bilinguals.

DETAILED DESCRIPTION:
Background:

Clinical observations and neuroimaging studies seem to confirm the role of executive functions and frontal structures in language processing in bilingual subjects.

Repetitive transcranial magnetic stimulation, such as for example theta burst stimulation (TBS), is increasingly being used as a valuable tool for neuroscientists investigating the underlying mechanisms of cognitive functions. Case studies have shown a change in language switching after bilingual patients received repetitive magnetic stimulation to the left DLPFC. However, there is no study investigating the effect of TBS applied to the DLPFC on language switching in healthy participants.

Procedure:

A planned total of 40 unbalanced bilingual participants will be included. Half of the participants will receive inhibitory theta burst stimulation (continuous TBS), the other half excitatory theta burst stimulation (intermittent TBS). After TBS, different language and nonverbal tasks will be performed while an EEG is measured. Before being stimulated, each subject will conduct the same tasks with a sham-TBS as a baseline measure.

ELIGIBILITY:
Inclusion Criteria:

* L1 (Swiss)German, knowledge of English as a foreign language
* 18-45 years of age
* right-handedness

Exclusion Criteria:

* epilepsy / family history of epilepsy
* brain surgery, traumatic brain injuries
* cardiac pacemaker, metallic objects in the head
* history of neurological diseases or severe psychiatric disorders
* drug use (alcohol, psychoactive medication)
* strong headache
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Annoni, Prof. Dr., Principal Investigator — University of Fribourg
Locations (1):
- Laboratory for Cognitive and Neurological Sciences, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holtzheimer P, Fawaz W, Wilson C, Avery D. Repetitive transcranial magnetic stimulation may induce language switching in bilingual patients. Brain Lang. 2005 Sep;94(3):274-7. doi: 10.1016/j.bandl.2005.01.003. PMID 16098377
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Nardone R, De Blasi P, Bergmann J, Caleri F, Tezzon F, Ladurner G, Golaszewski S, Trinka E. Theta burst stimulation of dorsolateral prefrontal cortex modulates pathological language switching: A case report. Neurosci Lett. 2011 Jan 10;487(3):378-82. doi: 10.1016/j.neulet.2010.10.060. Epub 2010 Oct 29. PMID 21036201

RESULTS

PARTICIPANT FLOW:
Groups:
- iTBS Group: intermittent theta burst stimulation (iTBS) + Sham iTBS
  * Sham iTBS: Placebo stimulation (3 Min)
  * Tasks (30 Min)
  * Pause (10Min)
  * iTBS: Excitatory stimulation (3Min)
  * Tasks (30Min)
- cTBS Group: continuous theta burst stimulation (cTBS) + Sham cTBS
  * Sham cTBS: Placebo stimulation (40Sec)
  * Tasks (30min)
  * Pause (10Min)
  * cTBS: inhibitory stimulation (40 Sec)
  * Tasks (30Min)
Period: Overall Study
Arm/Group | iTBS Group | cTBS Group
Started | 21 (21 Participants completed the Tasks following Sham-stimulation) | 20 (20 Participants completed the Tasks following Sham-stimulation)
Completed | 20 (20 Participants completed the Tasks following iTBS-stimulation) | 20 (20 Participants completed the Tasks following cTBS-stimulation)
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intermittent Theta Burst Stimulation: intermittent theta burst stimulation (iTBS) + Sham iTBS
  Sham iTBS: Placebo stimulation
  intermittent theta burst stimulation (iTBS): Excitatory rTMS
- Continuous Theta Burst Stimulation: continuous theta burst stimulation (cTBS) + Sham cTBS
  Sham cTBS: Placebo stimulation
  continuous theta burst stimulation (cTBS): inhibitory rTMS
- Total: Total of all reporting groups
Arm/Group | Intermittent Theta Burst Stimulation | Continuous Theta Burst Stimulation | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (2.7) | 22.8 (5.36) | 22.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: RTs for Picture Naming With the Factors Language (L1, L2) and Block (Switching, Non-Switching)
Description: Picture naming with the factors Language (L1, L2) and Block (Switching, Non-Switching): Speech onset times (msec) L1 refers to the mother tongue. L2 refers to the late acquired (> age 7) second language. Switching Block refers to a language switching block with picture naming alternated between the mother tongue and the second language.
  Non-Switching Block refers to a block of picture naming either only in the mother or only in the second language.
Time Frame: Within 30 minutes after intervention
Population: As a primary outcome we compared RTs following iTBS vs cTBS. Sham-TBS is only used to have a baseline control between the two groups
Measure: Mean (Standard Deviation); unit: Milliseconds
Groups:
- RTs for PN After Intermittent Theta Burst Stimulation: intermittent theta burst stimulation (iTBS) - across switching and non-switching blocks and across L1 and L2.
- RTs for PN After Continuous Theta Burst Stimulation: continuous theta burst stimulation (cTBS) - across switching and non-switching blocks and across L1 and L2.
- RTs for Picture Naming in L1: Voice onset times for Picture Naming in L1 - across switching and non-switching blocks and across iTBS and cTBS.
- RTs for Picture Naming in L2: Voice onset times for Picture Naming in L2 - across switching and non-switching blocks and across iTBS and cTBS.
- RTs for Picture Naming in the Non-switching Blocks: Voice onset times for Picture Naming in the non-switching blocks - across L1 and L2 and across iTBS and cTBS.
- RTs for Picture Naming in the Switching Blocks: Voice onset times for Picture Naming in the switching blocks - across L1 and L2 and across iTBS and cTBS.
Arm/Group | RTs for PN After Intermittent Theta Burst Stimulation | RTs for PN After Continuous Theta Burst Stimulation | RTs for Picture Naming in L1 | RTs for Picture Naming in L2 | RTs for Picture Naming in the Non-switching Blocks | RTs for Picture Naming in the Switching Blocks
Number analyzed (Participants) | 20 | 20 | 40 | 40 | 40 | 40
Milliseconds | 1103.32 (126) | 1107.26 (131) | 1098.82 (405) | 1158.91 (432) | 1081.14 (414) | 1175.24 (420)
Statistical Analysis 1: Comparison: RTs for PN After Intermittent Theta Burst Stimulation vs RTs for PN After Continuous Theta Burst Stimulation vs RTs for Picture Naming in L1 vs RTs for Picture Naming in L2 vs RTs for Picture Naming in the Non-switching Blocks vs RTs for Picture Naming in the Switching Blocks; Test type: Other; p = 0.932, Mixed Models Analysis — This p-value refers to the effect of stimulation (cTBS vs iTBS)

2. Secondary Outcome: Nonverbal Switching
Description: Nonverbal Switching: response times
Time Frame: Within 30 minutes after intervention
Population: Data are compared between iTBS and cTBS Sham-TBS is only used to have a baseline control between the two groups
Measure: Mean (Standard Deviation); unit: Milliseconds
Groups:
- Intermittent Theta Burst Stimulation: intermittent theta burst stimulation (iTBS)
- Continuous Theta Burst Stimulation: continuous theta burst stimulation (cTBS)
Arm/Group | Intermittent Theta Burst Stimulation | Continuous Theta Burst Stimulation
Number analyzed (Participants) | 20 | 20
Milliseconds | 772.07 (159.28) | 739.32 (137.23)
Statistical Analysis 1: Comparison: Intermittent Theta Burst Stimulation vs Continuous Theta Burst Stimulation; Test type: Other; p = 0.642, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 3 hours
Groups:
- cTBS: continuous theta burst stimulation (cTBS)
- iTBS: intermittent theta burst stimulation (iTBS)
- Sham iTBS: Placebo (baseline) stimulation for iTBS group
- Sham cTBS: Placebo (baseline) stimulation for cTBS group
Arm/Group | cTBS | iTBS | Sham iTBS | Sham cTBS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/21 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cTBS (N=20) | iTBS (N=20) | Sham iTBS (N=21) | Sham cTBS (N=20)
Nausea (Cardiac disorders) | 0 | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03148470/Prot_SAP_000.pdf